CLINICAL TRIAL: NCT06525831
Title: Multimodal Imaging of the Biomechanical Properties of Kidney Tumors: Feasibility, Inter-modality Correspondence and Diagnostic Value
Brief Title: Rein 3D PRINT MECHANICS
Acronym: Rein3DP-M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Sophia Genetics SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/11
Record Dates: First submitted 2024-07-11; First posted 2024-07-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Kidney Cancer
Keywords: Renal-Cell Carcinoma; Renal Elasticity; Biomarkers; Ultrasound; CT-scan; Magnetic Resonance Imaging; AFRI; Diffusion weighted imaging
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: The participants will undergo a Magnetic Resonance-elastography and Ultrasound exams for the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with kidney cancer surgery (Experimental): the patients will have an additionnal MRI elastography and Ultrasound exams for the research. The exams will be performed between the inclusion of the patient and the day before the surgery.
  Both exams are non-invasive, without radiation
  Interventions: Diagnostic Test: MR-elastography exam; Diagnostic Test: Ultrasound exam

INTERVENTIONS:
Diagnostic Test: MR-elastography exam — Imaging acquisition
Diagnostic Test: Ultrasound exam — Imaging acquisition

SUMMARY:
The goal of this innovative project is to evaluate the correspondence between several imaging modalities for characterizing the elasticity of healthy and pathological renal tissue which could help improve the realism of 3D prints used by urological surgeons and allow the identification of new, complementary imaging biomarkers. The main objective is to develop a predictive model of the biomechanical properties of normal and pathological kidney tissue, as assessed by the reference method (Magnetic Resonance (MR)-elastography).

DETAILED DESCRIPTION:
Medical imaging plays a key role in the diagnostic and therapeutic management of renal cell carcinomas. It can be used to confirm the presence of a tumor, localize it, suggest malignancy or even histological subtype, guide sampling, perform TNM staging, assist in surgical scheduling, monitor therapeutic efficacy in the event of systemic treatment, guide ablathermy procedures and look for relapses after curative treatments have ended. Imaging of kidney tumors relies on three complementary imaging modalities: ultrasound (US), Computed Tomography based on X-ray absorption (CT-scan) and magnetic resonance imaging (MRI). The most commonly performed examination remains the CT scan, which is used to print 3D models. However, the correlation between renal parenchyma densities and renal tumors (before and during the scan acquisition times after injection) and elasticity parameters measured by US and MRI has never been explored.

This trial aim to evaluate the correspondence between several imaging modalities for characterizing the elasticity of healthy and pathological kidney tissue. It will also improve the realism of 3D models used by surgeons, and identify new complementary imaging biomarkers.

To achieve this aim, 50 patients will undergo DWI -elastography (Diffusion Weigthed Imaging-elastography) and MR-elastography sequences, as well as an US before the surgery. After surgery, a fragment of the resected specimen will be used to perform mechanical tests to determine the real hardness of the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Scheduled for surgical management with nephrectomy for kidney tumor in the urology department of Bordeaux University Hospital
* CT scan available or scheduled for surgery
* Consent expressed for integration of the UroCCR database
* Expressed consent for participation in the Rein 3D Print Mechanics study
* Patients affiliated or benefiting from social security system

Exclusion Criteria:

* - Pregnant or breast-feeding women
* Contraindication to MRI (Magnetic Resonance Imaging)
* Contraindication to injection of gadoline contrast agents
* Biopsy prior to MRI, CT and ultrasound scans (risk of artifactual alteration, via iatrogenic hemorrhagic changes, of the biomechanical properties of the renal tumor and parenchyma).
* Presence of thoracolumbar arthrodesis material
* Obese patient (body mass index ≥ 30 kg/m²)
* Cystic renal tumors with solid component (corresponding to either parietal thickening or tumor bud) < 2 cm
* Necrotic renal tumors with solid component (corresponding to either parietal thickening or tumor bud) < 2 cm
* Ascites
* Person under legal protection
* Difficulty understanding and expressing in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-05-07 (Estimated); Study Completion 2027-05-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of the root mean square error (RMSE) | Between Day 0 and Month 4
  The aim is to successfully predict μMRE from dCT-, dCT40s, dCT90s, dCT10min (naming μCT the scan model prediction) with the lowest possible error.

SECONDARY OUTCOMES:
Measure of Spearman's rho | Between Day 0 and Month 4
  Researh of the highest possible value (maximum = 1).
Measure of the qualitative assessment | Between Day 0 and Month 4
  Measure based on a 5-point ordinal qualitative scale
Measure of the contrast | Between Day 0 and Month 4
  Calculation using the contrast-to-noise ratio
Measure of the noise | Between Day 0 and Month 4
  Calculation using the signal-to-noise ratio
Identification of imaging faisability limiting factors | Between Day 0 and Month 4
  Evaluation of the number of situations where the examination has no clinical diagnostic value and associations with potential limiting factors by using a composite criteria including :
  * body mass index
  * sarcopenia,
  * lesion location
  * lesion size
  * lesion architecture
Evaluation of imaging repetabiliy limiting factors | Between Day 0 and Month 4
  Measurement of the intra-class correlation coefficients and Bland-Altmann plot traces.
  The aim is for the intra-class score to be as high as possible (maximum = 1, ideally >0.90).
identification of decorrelation situations and potential bias between biomechanical properties obtained by hardness measurements in the different imaging modalities | Between Day 0 and Month 4
  Visual measurement for each patient and anatomical situation with possible matching, point clouds with in X the hardness obtained by one imaging modality and in Y the hardness obtained by another imaging modality. The descriptive characteristics of the points (voxel or patient segmentation) with decorrelation will then be analyzed.
Carry out associations between histological categorical variables and numerical elasticity variables | Between Day 0 and Month 4
  The measurement will be based on associations between categorical histological and numerical elasticity variables, with area under the ROC curve comparisons or cut-off identification where appropriate.
  Malignant/benign character (binary variable) and histological type (non- ordinal categorical variable) will be assessed as part of routine care by the pathologist.
Verification of correlation between actual hardness and hardness assessed by the various imaging methods, carried out directly on a fragment of the fresh surgical specimen | Between Day 0 and Month 4
  The actual hardness in kPa will be assessed by the physician in the immediate post-operative period on the fragment of the fresh surgical specimen, using a destructive method which measures a tissue's resistance to compression. The tissue will be subjected to increasing compression until it breaks.
  The value wil be compared with data obtained by imaging.

CONTACTS AND LOCATIONS:
Overall Officials: JAMBON EVA, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France